CLINICAL TRIAL: NCT05843331
Title: Vertical Implant Versus Inclined Implant to Retain Locator Maxillary Overdenture : One Year Randomized Controlled Clinical Trial
Brief Title: Vertical Versus Inclined Implant to Retain Locator Maxillary Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A26060722
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Implant Complication; Bone Loss
Keywords: maxillary overdentures; angled abutment; locator
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial study conducted on 12 participants with completely edentulous maxillary ridges. Patients were allocated into one of two treatment groups: 1) The control group ; included 6 patients (3 males and 3 females) who will receive 4 vertical implants with straight trans mucosal abutments retaining locator maxillary overdenture 2) The study group; include 6 participants (3 males and 3 females) who will receive 4 inclined implants with angled trans mucosal abutments for retaining locator maxillary overdenture. A new maxillary conventional dentures will be constructed with a bilateral balanced occlusal concept for all patients. Maxillary dentures were duplicated into heat cure acrylic resin dentures to be used as a radiographic template. Four implants were inserted in the maxilla . For both groups, locator abutments were screwed to the abutments .Clinical and radiographic evaluations were done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posterior vertical implants (Active Comparator): the anterior implants were inserted in the canine/lateral incisor area bilaterally to each other's following the contour of the alveolar bone of the premaxilla. The posterior implants were inserted vertically just anterior to the maxillary sinus (in the area of second premolars) .
  Interventions: Procedure: implants
- posterior inclined implants (Active Comparator): The anterior implants were inserted in the canine/lateral incisor area bilaterally to each other's and will be inclined 15o labially following the contour of the alveolar bone of the premaxilla. The posterior implants were inserted just anterior to the maxillary sinus (in the area of second premolars) and inclined 15o distally .
  Interventions: Procedure: implants

INTERVENTIONS:
Procedure: implants — Four implants in the maxilla with locator attachments

SUMMARY:
Objectives: evaluate the success rate, prosthetic maintenance , clinical and radiologic results of vertical implants with straight abutments versus inclined implants with angled abutments to retain locator maxillary overdentures. There were two groups : 1) The control group 2) The study group

DETAILED DESCRIPTION:
the aim of the present investigation was to evaluate the success rate, prosthetic maintenance , clinical and radiologic results of vertical implants with straight abutments versus inclined implants with angled abutments to retain locator maxillary overdentures.

Materials and Methods conducted on 12 patients (6 males and 6 females) aged 58 to 68 years with completely edentulous maxillary ridges opposing implant-retained mandibular overdentures. Patients admit to the prosthodontic department, Faculty of Dentistry, Mansoura University for oral rehabilitation by implant-supported maxillary prostheses. Patients were allocated into one of two treatment groups: 1) The control group ; included 6 patients (3 males and 3 females) who will receive 4 vertical implants with straight trans mucosal abutments retaining locator maxillary overdenture 2) The study group; include 6 patients (3 males and 3 females) who will receive 4 inclined implants with angled trans mucosal abutments for retaining locator maxillary overdenture. Randomization and allocation of patients into treatment groups was made by dental personnel who is blind to treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Unable to wear the upper denture
2. Radiographic diagnosis of bone loss

Exclusion Criteria:

1. Neuromuscular diseases
2. Insulin dependent diabetes

Ages: 58 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 6 males and 6 females
Enrollment: 12 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
plaque index | 12 months
  measure plaque around each implant using Mombelli indices
pocket depth | 12 months
  dental probe used to measure the depth of formed pocket around each implant
implant stability | 12 months
  stability of each implant measured using Osstell® device

SECONDARY OUTCOMES:
Radiographic outcome | 12 months
  measuring bone resorption using the long-cone standardized periapical radiography

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Aboelez, Phd, Principal Investigator — Mansoura University; Mostafa Elsyad, Phd, Study Chair — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ELsyad MA, Emera RM, Ashmawy TM. Effect of Distal Implant Inclination on Dislodging Forces of Different Locator Attachments Used for Mandibular Overdentures: An In Vitro Study. J Prosthodont. 2019 Feb;28(2):e666-e674. doi: 10.1111/jopr.12710. Epub 2017 Nov 16. PMID 29143403
- [Background] ELsyad MA, Abo Hatem OE, Shawky AF, Emera RMK. Effect of Different Degrees of Mesial Implant Inclination on the Retention and Stability of Two-Implant Mandibular Overdentures Retained with Stud Attachments: An In Vitro Study. Int J Oral Maxillofac Implants. 2018 March/April;33(2):259-268. doi: 10.11607/jomi.5791. Epub 2017 Oct 13. PMID 29028850